CLINICAL TRIAL: NCT07295353
Title: Accelerating Recovery After ICU Admission: Post-discharge Supplementation With Pasteurized Akkermansia Muciniphila.
Acronym: PAM-ICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: THE AKKERMANSIA COMPANY (Unknown); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, W. J. Wiersinga, MD, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL-009844
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; Post Intensive Care Unit Syndrome; Critical Illness; Microbiome Dysbiosis; Intensive Care Unit Survivors
Keywords: Pasteurized Akkermansia muciniphila; Akkermansia muciniphila; Postbioticum; Microbiome; PAM; Gut Barrier Function; Post-Sepsis Recovery; Randomized Controlled Trial
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a parallel-group design to receive either pasteurized Akkermansia muciniphila supplementation or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, placebo-controlled trial. Participants, care providers, investigators, and outcomes assessors are masked to intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pasteurized Akkermansia muciniphila (PAM) (Experimental): Oral supplementation with pasteurized Akkermansia muciniphila, 30 × 10⁹ bacteria in capsule form, once daily for 56 days, in addition to standard care.
  Interventions: Dietary Supplement: Pasteurized Akkermansia muciniphila
- Placebo (Placebo Comparator): Oral administration of placebo capsules matched in appearance and dosing schedule to the PAM capsules, once daily for 56 days, in addition to standard care. The placebo contains no active component.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Dietary Supplement: Pasteurized Akkermansia muciniphila — Oral supplementation with pasteurized Akkermansia muciniphila, 30 × 10⁹ bacteria in capsule form, once daily for 56 days, in addition to standard care.
  Arms: Pasteurized Akkermansia muciniphila (PAM)
Other: Placebo Control — Oral administration of placebo capsules matched in appearance and dosing schedule to the PAM capsules, once daily for 56 days, in addition to standard care. The placebo contains no active component.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if daily oral supplementation with pasteurized Akkermansia muciniphila (PAM), an EFSA-approved food supplement, can support recovery in adults who have recently been treated in the ICU for sepsis.

The main questions it aims to answer are:

* Is PAM safe to take for 56 days after ICU discharge?
* Does PAM increase the abundance of beneficial butyrate-producing bacteria in the gut?

Researchers will compare PAM to a placebo (a capsule that looks the same but has no active ingredient) to see if PAM improves gut microbiota and immune recovery.

Participants will:

* Take PAM or placebo capsules once daily for 56 days
* Provide stool and blood samples at baseline, day 28, and day 56
* Receive a follow-up phone call about their health 1 year after starting the study

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Treated in the ICU for at least 2 days and discharged to a regular clinical ward
* Diagnosed with sepsis during ICU admission
* Received selective digestive decontamination (SDD) or cephalosporin
* Capable of giving written informed consent

Exclusion Criteria:

* Recent major gastrointestinal surgery
* Diagnosed with ulcerative colitis or Crohn's disease
* Presence of a hematological malignancy and/or current use of immunomodulatory therapy (e.g., CAR-T cell therapy or immune checkpoint inhibitors) Use of systemic immunomodulatory drugs or corticosteroids (defined as ≥10 mg prednisone equivalent daily at ICU discharge), at the time of inclusion.
* History of solid organ or stem cell transplantation
* Pregnancy or lactation
* Donation of blood or plasma within 30 days prior to inclusion or planned donation during the intervention period
* Any other condition that, in the opinion of the investigator, could pose a risk to the subject or interfere with study result

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in abundance of butyrate-producing bacteria | Baseline and day 56
  Difference (Δ) from baseline in the relative abundance of gut butyrate-producing bacteria at day 56, assessed by shotgun metagenomic sequencing (taxa/functional pathways associated with butyrate production), comparing PAM vs placebo at the end of the intervention
Safety (occurrence of adverse events) | Baseline to day 56 (end of intervention)
  Proportion of participants with ≥1 adverse event (AE) and total AE count, summarized by severity and relatedness, comparing PAM vs placebo at end of intervention

SECONDARY OUTCOMES:
Changes in gut microbiota composition | Day 0 (baseline), day 28, day 56
  Differences between arms and within-participant change from baseline in microbiota α-diversity and β-diversity
Changes in circulating immune and inflammatory profiles | Day 0 (baseline), day 28, day 56
  Between-arm differences and longitudinal changes in systemic immune profiles, including major innate and adaptive subsets and activation markers. In addition, ex vivo whole blood stimulations will be performed to quantify cytokine production in response to microbial ligands.
Changes in gut barrier markers | Day 0 (baseline), day 28, day 56
  Plasma levels and changes from baseline of lipopolysaccharide-binding protein (LBP) and soluble CD14 (sCD14); between-arm comparisons.
Secondary infections and rehospitalizations | Through day 365
  Incidence of adjudicated secondary infections and all-cause rehospitalizations; comparison between PAM and placebo.

OTHER OUTCOMES:
Host metabolic function | Day 0 (baseline), day 28, day 56
  Change from baseline in insulin sensitivity estimated by HOMA-%S, calculated from fasting plasma glucose and insulin; between-arm differences.

CONTACTS AND LOCATIONS:
Overall Officials: JW Wiersinga, Professor, Principal Investigator — Amsterdam UMC

IPD SHARING:
Plan to Share IPD: No